CLINICAL TRIAL: NCT03493828
Title: A Randomized Double Blinded Controlled Trial on the Efficacy of TAP Block in Cesarean Section Patients When Compared to Placebo
Brief Title: Efficacy of TAP Block in Cesarean Section Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Joel Yarmush, MD, New York Presbyterian Brooklyn Methodist Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAP2013
Record Dates: First submitted 2015-04-27; First posted 2018-04-11 (Actual); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Pain Control
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Arm 1: Bupivacaine 05%, arm 2: Bupivacaine 0.25%, and arm 3: placebo (Normal saline)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization sheet was given to someone who is not involved in the study, also the person who prepare the medicine is not involved in the study.
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAP using Bupivacaine 0.5% (Active Comparator): Following completion of the Cesarean delivery, the abdomen was aseptically prepped with ChloraPrep®. A Sonosite ultrasound machine (S-nerve) with a 14-8 MHz linear probe was used to visualize the lateral abdominal wall muscles and transversus abdominis plane. A 2 or 4 inch stimuplex (Braun) needle was advanced under ultrasound guidance to the transversus abdominis plane. After negative aspiration, 15 ml of Bupivacaine 0.5% was incrementally injected on each side. The spread of solution within the transversus abdominis plane was visualized with the ultrasound.
  Interventions: Procedure: TAP block using Bupivacaine 0.5%
- TAP using Bupivacaine 0.25% (Active Comparator): Following completion of the Cesarean delivery, the abdomen was aseptically prepped with ChloraPrep®. A Sonosite ultrasound machine (S-nerve) with a 14-8 MHz linear probe was used to visualize the lateral abdominal wall muscles and transversus abdominis plane. A 2 or 4 inch stimuplex (Braun) needle was advanced under ultrasound guidance to the transversus abdominis plane. After negative aspiration, 15 ml of Bupivacaine 0.25% was incrementally injected on each side. The spread of solution within the transversus abdominis plane was visualized with the ultrasound.
  Interventions: Procedure: TAP block using Bupivacaine 0.25%
- Placebo (Placebo Comparator): Following completion of the Cesarean delivery, the abdomen was aseptically prepped with ChloraPrep®. A Sonosite ultrasound machine (S-nerve) with a 14-8 MHz linear probe was used to visualize the lateral abdominal wall muscles and transversus abdominis plane. A 2 or 4 inch stimuplex (Braun) needle was advanced under ultrasound guidance to the transversus abdominis plane. After negative aspiration, 15 ml of normal saline was incrementally injected on each side. The spread of solution within the transversus abdominis plane was visualized with the ultrasound.
  Interventions: Procedure: TAP block using Normal Saline

INTERVENTIONS:
Procedure: TAP block using Bupivacaine 0.5% — Following completion of the Cesarean delivery, the abdomen was aseptically prepped with ChloraPrep®. A Sonosite ultrasound machine (S-nerve) with a 14-8 MHz linear probe was used to visualize the lateral abdominal wall muscles and transversus abdominis plane. A 2 or 4 inch stimuplex (Braun) needle was advanced under ultrasound guidance to the transversus abdominis plane. After negative aspiration, 15 ml of Bupivacaine 0.5% was incrementally injected on each side. The spread of solution within the transversus abdominis plane was visualized with the ultrasound.
  Arms: TAP using Bupivacaine 0.5%
Procedure: TAP block using Bupivacaine 0.25% — Following completion of the Cesarean delivery, the abdomen was aseptically prepped with ChloraPrep®. A Sonosite ultrasound machine (S-nerve) with a 14-8 MHz linear probe was used to visualize the lateral abdominal wall muscles and transversus abdominis plane. A 2 or 4 inch stimuplex (Braun) needle was advanced under ultrasound guidance to the transversus abdominis plane. After negative aspiration, 15 ml of Bupivacaine 0.25% was incrementally injected on each side. The spread of solution within the transversus abdominis plane was visualized with the ultrasound.
  Arms: TAP using Bupivacaine 0.25%
Procedure: TAP block using Normal Saline — Following completion of the Cesarean delivery, the abdomen was aseptically prepped with ChloraPrep®. A Sonosite ultrasound machine (S-nerve) with a 14-8 MHz linear probe was used to visualize the lateral abdominal wall muscles and transversus abdominis plane. A 2 or 4 inch stimuplex (Braun) needle was advanced under ultrasound guidance to the transversus abdominis plane. After negative aspiration, 15 ml of normal saline was incrementally injected on each side. The spread of solution within the transversus abdominis plane was visualized with the ultrasound.
  Arms: Placebo

SUMMARY:
TAP Block done with 2 different concentrations of bupivacaine and placebo

DETAILED DESCRIPTION:
TAP Block was done using 2 different concentrations of bupivacaine (0.5% and 0.25%) and placebo and the post operative sedation was measured in each arm and compared together.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women

Exclusion Criteria:

* Allergy to local anesthetics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adel Guirguis, MD, MS, Study Director — New York Presbyterian Brooklyn Methodist Hospital
Locations (1):
- New York Methodist Hospital, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAP Using Bupivacaine 0.5% | TAP Using Bupivacaine 0.25% | Placebo
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP Using Bupivacaine 0.5% | TAP Using Bupivacaine 0.25% | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 33 [23 to 41] | 34.5 [21 to 48] | 32.5 [19 to 41] | 33 [19 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 20 | 60
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  North America | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Effect of Transversus Abdominis Plane (TAP) Block Using Either 0.5% or 0.25% Bupivacaine on Analgesia for Cesarean Section Patients When Compared to Placebo.
Description: The total the number of Patient Controlled Analgesia (PCA) boluses used by the patients postoperatively within 24 hours
Time Frame: 0-24 hours
Population: Number of PCA bolus used within 24 hours
Measure: Mean (Standard Error); unit: PCA bolus
Arm/Group | TAP Using Bupivacaine 0.5% | TAP Using Bupivacaine 0.25% | Placebo
Number analyzed (Participants) | 20 | 20 | 20
PCA bolus | 9.45 (1.292) | 8.95 (1.756) | 17.65 (2.893)

ADVERSE EVENTS:
Time Frame: Within 72 hours post operatively.
Arm/Group | TAP Using Bupivacaine 0.5% | TAP Using Bupivacaine 0.25% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
The investigators used epidural morphine in all 3 groups, so they were unable to assess whether TAP block in a multimodal analgesic regimen without the neuraxial opioids provide advantage over the multimodal analgesic regimen with neuraxial opioids.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes